CLINICAL TRIAL: NCT05384756
Title: A Pilot Study of Nonmyeloablative Regimen Using Total Marrow and Lymphoid Irradiation for Irradiation Sparing of Bystander Organs in Hematopoietic Cell Transplantation From Matched Related or Unrelated Donor in Patients With Sickle Cell Disease
Brief Title: TMLI and Alemtuzumab for Treatment of Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20682; NCI-2022-03571 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20682 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Radiotherapy, Intensity-Modulated; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TMLI, alemtuzumab) (Experimental): Patients receive alemtuzumab IV over 4 hours QD on days -7 to -3. Patients undergo TMLI BID on day -2. Patients also undergo HCT on day 0 and receive sirolimus on day -1 and day 0.
  Interventions: Drug: Alemtuzumab; Procedure: Hematopoietic Cell Transplantation; Radiation: Intensity-Modulated Radiation Therapy; Drug: Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab — Given IV
  Other Names: Anti-CD52 Monoclonal Antibody; Campath; Campath-1H; LDP-03; Lemtrada; MabCampath; Monoclonal Antibody Campath-1H
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Radiation: Intensity-Modulated Radiation Therapy — Undergo TMLI
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Sirolimus — Medication to prevent the development of graft-versus-host disease (GVHD)
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217

SUMMARY:
This phase I trial tests the safety and effectiveness of total marrow and lymphoid irradiation (TMLI) and alemtuzumab as a conditioning regimen in patients with sickle cell disease. Conditioning regimens are treatments used to prepare a patient for stem cell transplantation. A stem cell transplant is a procedure in which a person receives blood stem cells, which make any type of blood cell. A conditioning regimen may include chemotherapy, monoclonal antibody therapy, and radiation to the entire body. It helps make room in the patient's bone marrow for new blood stem cells to grow, and helps prevent the patient's body from rejecting the transplanted cells. Alemtuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Graft-versus-host disease (GVHD) is a complication that may occur after hematopoietic cell transplantation (HCT) in which donated cells view the recipient's cells as foreign and attack them. Giving TMLI and alemtuzumab may help reduce organ damage that can be caused by radiation and decrease the risk of GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and feasibility of a fixed TMLI dose of 600 cGy with alemtuzumab as non-myeloablative conditioning (NMC) regimen in patients with sickle cell disease to achieve stable engraftment by Day +100 post HCT.

SECONDARY OBJECTIVES:

I. Assess the hematopoietic recovery by determining donor neutrophil engraftment, platelet engraftment.

II. Assess irradiation doses to non-target organs (lungs, heart, liver, spleen, kidneys, and gonads).

III. Assess the incidence of acute GvHD (grade II - IV) during the first 100 days after transplantation and chronic GvHD at 1 year post-HCT.

IV. Assess overall, event-free, and disease free survival at 1 year post-HCT. V. Assess donor chimerism at day +100 and 1 and 2 years after HCT.

EXPLORATORY OBJECTIVES:

I. Assess immune reconstitution post HCT on baseline, then on days +15, +30, +60, and +180, and 1-year post-HCT. II. Assessment of quality of life at baseline, Day+100, Day +180 and at 1-year post-HCT.

III. Define the impact of sickle cell disease (SCD) including inflammation on the bone marrow microenvironment and hematopoietic cells function at baseline.

IV. Monitor treatment response noninvasively on the recovery of bone marrow microenvironment (hematopoietic and vascular).

V. Monitor treatment response noninvasively on cerebral blood flow (CBF).

OUTLINE:

Patients receive alemtuzumab intravenously (IV) over 4 hours once daily (QD) on days -7 to -3. Patients undergo TMLI twice daily (BID) on day -2. Patients also undergo HCT on day 0 and receive sirolimus on day -1 and day 0.

After study treatment, patients are followed up on day 30, and for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Registered into Risk Evaluation and Mitigation Strategies (REMS) program
* Age: 12-40 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Have a diagnosis of sickle cell disease, be at a high risk for disease related morbidity or mortality, which must be defined by one of the following disease status criteria:

  * Significant neurologic event (stroke) or any neurological deficit lasting > 24 hours; or increased transcranial Doppler velocity (> 200 m/s).
  * History of one or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea).
  * History of one or more severe vaso-occlusive pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea).
  * Recurrent priapism requiring medical therapy.
  * Osteonecrosis of two or more joints despite the institution of supportive care measures.
  * Prior treatment with regular red blood cell (RBC) transfusion therapy, defined as receiving 8 or more transfusions per year for > 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
  * Echocardiograph finding of tricuspid valve regurgitation jet (TRJ) velocity >= 2.5 m/sec.
* Have a related donor who is matched on at least 8/10 human leukocyte antigen (HLA)-A, B, C, and DRB1 Loci
* Total bilirubin =< 2.5 x upper limit normal (ULN( (unless has Gilbert's disease) (performed within 30 days prior to day 1 of protocol)
* Aspartate aminotransferase (AST) =< 1.5 x ULN (performed within 30 days prior to day 1 of protocol)
* Alanine aminotransferase (ALT) =< 1.5 x ULN (performed within 30 days prior to day 1 of protocol)
* Creatinine clearance (CrCl) of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 30 days prior to day 1 of protocol)
* If not receiving anticoagulants: International Normalized Ratio (INR) OR Prothrombin (PT) =< 1.5 x ULN (performed within 30 days prior to day 1 of protocol)

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated Partial Thromboplastin Time (aPTT) =<1.5 x ULN (performed within 30 days prior to day 1 of protocol)

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Left ventricular ejection fraction (LVEF) >= 50% (performed within 30 days prior to day 1 of protocol)

  * Note: To be performed within 28 days prior to Day 1 of protocol therapy.
* If able to perform pulmonary function tests: Forced expiratory volume in 1 second (FEV1), force vital capacity (FVC), and diffused lung capacity of carbon monoxide (DLCO) (diffusion capacity) >= 50% of predicted (corrected for hemoglobin)

  * If unable to perform pulmonary function tests: Oxygen (O 2) saturation > 92% on room air
  * Note: To be performed within 28 days prior to Day 1 of protocol therapy.
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma regain [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be require.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least Six months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* DONOR: Age =< 60 years
* DONOR: Medical history and physical examination confirm good health status as defined by institutional standards
* DONOR: Serologies for: Hepatitis B (HBV) Core Antibody, HIV I/II Antibody, human T-lymphotropic virus (HTLV) - I/II antibody, HCV antibody, Hepatitis B surface antigen, Serologic Test for Syphilis, HIV-1/HCV/HBV nucleic acid, West Nile virus nucleic acid, Trypanosoma cruzi antibody, Cytomegalovirus (CMV) antibody, (AKA: Donor Room Serologies)
* DONOR: Female donors of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (b-HCG) test within 30 days of initiation of conditioning, 30 days of patients admission for conditioning and 7 days of mobilization or bone marrow harvest.
* DONOR: The donor must be informed of the investigational nature of this study and have signed a consent form in accordance with Federal Guidelines and the guidelines of the participating institution

Exclusion Criteria:

* Prior allogeneic or autologous stem cell transplant
* Patients who are receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.
* History of allergic reactions attributable to compounds of similar chemical or biologic composition to study agent
* Patients with any active malignancy are ineligible for this study, other than non-melanoma skin cancers
* Medical problem or neurologic/psychiatric dysfunction which would impair patient ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery which in the opinion of the principal investigator would place the recipient at unacceptable risk.
* Active infection requiring antibiotics
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* DONOR: Evidence of active infection
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis if donating peripheral stem cells or unlikely to tolerate general anesthesia and bone marrow collection if donating a bone marrow
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or granulocyte colony-stimulating Factor (G-CSF) therapy if donating peripheral stem cells or general anesthesia and bone marrow collection if donating a bone marrow
* DONOR: Lactating female or, if of child-bearing potential, is unwilling to implement adequate birth control
* DONOR: HIV positive
* DONOR: Prior radiation therapy

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day 100 post-transplant
  Will be scored on the Bearman Scale National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with the unacceptable adverse events will be calculated along with the appropriate Clopper-Pearson 90% confidence intervals.
Feasibility | Up to 2 years
  Feasibility will be defined as engraftment that would be sufficient to reduce sickle cell disease (SCD) burden (Any donor chimerism with Hgb S =< 30%).

SECONDARY OUTCOMES:
Platelet engraftment | Up to 2 years
  Platelet engraftment will be defined as independence from platelet transfusion for at least 7 days with a platelet count of more than >20 × 10^9/L
Time to acute graft-versus-host disease (grades 2-4 and 3-4) until day +100 after transplant | Up to 2 years
  Acute Graft versus Host Disease (aGVHD) of grades 2-4 and 3-4: Documented/biopsy proven acute graft versus host disease is graded according to the Consensus Grading. Time to event is measured from date of stem cell infusion to document/biopsy proven acute GVHD onset date (within the first 100 days post-transplant) and will be used to estimate the cumulative incidence.
Time to chronic graft-versus-host disease for up to one year after transplant | Up to 2 years
  Chronic Graft versus Host Disease (cGVHD): chronic Graft versus Host Disease (aGVHD) of grades 2-4 and 3-4:
  Documented/biopsy proven chronic graft versus host disease is scored according to NIH Consensus Staging. Time to event is measured from date of stem cell infusion to the documented/biopsy proven chronic GVHD onset date and will be used to estimate the cumulative incidence.
Overall survival (OS) | From start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 2 years
  Patients are considered a failure for this endpoint if they die, regardless of cause.
Event-free survival (EFS) | From start of protocol therapy to death, graft failure, or last follow-up, whichever comes first, assessed up to 2 years
  Patients are considered a failure for this endpoint if they graft failure, or die, regardless of cause. Time to this event is the time from start of protocol therapy to death, graft failure, or last follow-up, whichever comes first.
Disease-free Survival (DFS) | From date of stem cell infusion to death, disease relapse/progression, or last follow-up, whichever comes first, assessed up to 2 years
  Patients are considered a failure for this endpoint if they die (regardless of cause) or experience disease progression or relapse.

OTHER OUTCOMES:
Immune cell reconstitution | Up to 2 years
  Immune cell reconstitution will be assessed by flow cytometry analysis
Quality of life - PedsQL | Up to 2 years
  Items on the PedsQL Generic Core Scales are reverse scored and transformed to a 0-100 scale.
  Higher scores indicate better health related quality of life:
  0 ("Never") = 100
  1. ("Almost Never") = 75
  2. ("Sometimes") = 50
  3. ("Often") = 25
  4. ("Almost Always") = 0
  For adults 16-item QOLS patients will be given a copy of the 7-point response scale ["delighted" (7), "pleased" (6), "mostly satisfied" (5), "mixed" (4), "mostly dissatisfied" (3), "unhappy" (2), "terrible" (1).] The QOLS scores will be summed so that a higher score indicates higher quality of life. Average total score for healthy populations is about 90. However, like many QOL instruments, the means tend to be quite negatively skewed with most patients reporting some degree of satisfaction with most domains of their lives.
Bone marrow environment inflation - levels of inflammatory cytokines | Baseline only (pre-conditioning)
  The long-term impact of Sickle Cell Disease on patients bone marrow will be measured by evaluation of the levels of inflammatory cytokines in the bone marrow before treatment with TMLI and alemtuzumab.
Bone marrow environment inflation - stem cell function | Baseline only (pre-conditioning)
  The long-term impact of Sickle Cell Disease on patients bone marrow will be measured by evaluation of the stem cell function in the bone marrow before treatment with TMLI and alemtuzumab.
Treatment response on bone marrow environment and CBF | Up to 1 year
  Treatment response on bone marrow environment and CBF will be assessed by Computed Tomography (CT) and Magnetic Resonance Imaging (MRI). All imaging will be performed before the start of the treatment and post-transplant at days 30, 100, 180, and at one year, coinciding with time points when clinical standard biopsy samples are obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States